CLINICAL TRIAL: NCT01421680
Title: A Prospective Randomized Controlled Trial Evaluating the Effects of Preoperative and Postoperative Oral Nutritional Supplements (ONS) in Malnourished Post-gastrectomy Patients
Brief Title: The Effects of Preoperative and Postoperative Oral Nutritional Supplements in Malnourished Post-gastrectomy Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Han-Kwang Yang, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ANSK1101
Record Dates: First submitted 2011-08-17; First posted 2011-08-23 (Estimated); Last update posted 2014-03-14 (Estimated); Status verified 2014-03

CONDITIONS: Malnourished; Stomach Neoplasms; Gastrointestinal Stromal Tumors
MeSH Terms: conditions — Malnutrition; Stomach Neoplasms; Gastrointestinal Stromal Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ensure powder (Active Comparator): Oral Nutritional Supplements with carbohydrate, lipid, protein, vitamin and minerals
  Interventions: Dietary Supplement: Ensure powder
- Standard care (No Intervention): Standard care without oral nutritional supplements

INTERVENTIONS:
Dietary Supplement: Ensure powder — Ensure powder(500kcal) per day for 7 weeks
  Other Names: Ensure powder (Abbott)
  Arms: Ensure powder

SUMMARY:
The objective of this study is to evaluate the effect of a perioperative nutrition strategy using oral nutritional supplements (ONS) on postoperative complications and improvement in body weight in malnourished patients who underwent gastrectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 20 years
* Patients who undergo distal, total, proximal, or pylorus-preserving gastrectomy
* Patients who are assessed as moderate or severe malnourished according to PG-SGA or patients with BMI lower than 18.5 kg/m2
* Patients who can take oral meals
* Patients who agree on the informed consent

Exclusion Criteria:

* Emergent operation
* Patients who received preoperative chemotherapy or radiation therapy within 6 months
* Pregnant patients
* Patients who cannot consume the Ensure powder
* Patients who enrolled another clinical trials

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2011-08; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Postoperative complication rate | 7weeks

SECONDARY OUTCOMES:
Body weight | 7weeks
Body composition indices | 7weeks
Length of hospital stay | 7weeks
Quality of life | 7weeks
Postoperative 30-day mortality | 7weeks
Biochemical assessment of nutritional status | 7weeks
Readmission rate | 7weeks
Patient compliance of oral nutritional supplements | 7weeks

CONTACTS AND LOCATIONS:
Overall Officials: Han-Kwang Yang, M.D., Principal Investigator — Department of Surgery, Seoul National University Hospital
Locations (1):
- Department of Surgery, Seoul National University Hospital, Seoul, South Korea